CLINICAL TRIAL: NCT01888536
Title: A Randomized, Double-Blind, Comparative, Multi-Center, Phase Ⅳ Clinical Trial to Evaluate Efficacy of 『Opast Tablet』for Neurologic Claudication in Patients With Lumbar Spinal Stenosis
Brief Title: A Study to Evaluate Efficacy of 『Opast Tablet』for Neurologic Claudication in Patients With Lumbar Spinal Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YJ7-401
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Neurologic Claudication in Patients With Lumbar Spinal Stenosis
MeSH Terms: interventions — limaprost; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Limaprost & Placebo (Experimental): Limaprost 5㎍ tablet and a capsule of Pegabalin-Placebo thrice a day for 8 weeks.
  Interventions: Drug: Limaprost; Drug: Placebo(for Pregabalin)
- Pregabalin & Placebo (Active Comparator): Pregabalin 75mg capsule and a tablet of Limaprost-Placebo thrice a day for 8 weeks.
  Interventions: Drug: Pregabalin; Drug: Placebo(for Limaprost)
- Limaprost+Pregabalin (Active Comparator): Limaprost 5㎍ tablet and Pregabalin 75mg capsule thrice a day for 8 weeks.
  Interventions: Drug: Limaprost; Drug: Pregabalin

INTERVENTIONS:
Drug: Limaprost
  Other Names: Opast tablet
  Arms: Limaprost & Placebo; Limaprost+Pregabalin
Drug: Pregabalin
  Other Names: Rikalin capsule 75mg
  Arms: Limaprost+Pregabalin; Pregabalin & Placebo
Drug: Placebo(for Pregabalin) — mimic Pregabalin 75mg capsule
  Arms: Limaprost & Placebo
Drug: Placebo(for Limaprost) — mimic Limaprost tablet
  Arms: Pregabalin & Placebo

SUMMARY:
This trial is a comparative study of Opast tablet and Rikalin capsule 75mg and Rikalin capsule 75mg in combination with Opast tablet to evaluate improvement effectiveness of Opast tablet on subjective symptoms and neurologic claudication in patients with lumbar spinal stenosis.

DETAILED DESCRIPTION:
Subjects who provided written consents voluntarily after receiving a sufficient explanation about this trial will be assigned to one of groups(study group; limaprost, comparative group 1; pregabalin, comparative group 2; limaprost+ pregabalin) by randomization at the rate of 1:1:1.

Subjects will take assigned investigational drugs thrice a day for eight weeks by double-blind and double-dummy methods, and they will visit the site two times at intervals of four weeks.

At each site visit point, the improvement effectiveness will be comparatively evaluated by evaluation of following endpoints;

Efficacy endpoints: ICD(initial claudication distance) at treadmill test (speed:3km/hr, grade:0%), VAS in pain on lower extremities, EQ-5D and ODI Safety endpoints: Vital signs, hematology/blood chemistry tests and adverse events, etc.

ELIGIBILITY:
Inclusion Criteria:

* Subject is fully understand the clinical trial and obtained informed consent.
* Age 20-75years.
* Patients with a confirmed diagnosis of waist of spinal canal stenosis.
* Limb pain caused by waist of spinal canal stenosis index of VAS 3 or more patients.
* Subject who has numbness symptom on lower extremity(ies) and intermittent claudication that are due to spinal canal stenosis and fulfills both of following criteria at the same time

  * When screening visit, a medical examination by interview had the following symptoms in subjects ; In daily life walking, when walked by within 20 minutes on flatland, the subject can feel the symptoms (numbness, pain or tightness on lower extremity(ies), etc.)

    * Subject who experienced numbness, pain, tightness or other similar symptom(s) on lower extremity within 15 minutes from test start at baseline(D1) evaluation.

      * speed: 3km/hr, grade:0%, posture: should keep their lumbar spinal extended

Exclusion Criteria:

* Pregnant or lactating women of childbearing potential not employing adequate contraception.
* Patients who have the hereditary problem of galactose intolerance, Lapp lactase deficiency or grape sugar-galactose absorption defect.
* Patients with systemic disease affecting the lower limbs.
* Patients who have cauda equina syndrome.
* Patients with acute osteoporosis compression fracture in lumbar vertebra.
* Patients who have gait disturbance of degenerative arthritis by hip joint, knee joint, ankle joint.
* At least one month before the start of the study, patients use of steroid drug except lumbar dura mater.
* 6 month before the start of the study, patients with ischaemic disease in blood vessel, lung or the coronary artery, varicose artery.
* Patients with lumbar necrosis in head of femur avascular necrosis, necrotic foot ulcer.
* Patients surgery by lumbar fusion and lumbar decompression.
* Patients with renal disease or need to hemodialysis.

  * serum creatinine > 2xUNL
* 3 month before the start of the study, patients participated in another clinical research.
* Patients with difficult understanding spirit incompetence, lack of will or language barrier.
* The investigator judged seriously ill patients need surgery patient.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
baseline-adjusted Oswestry Disability Index score at 8 weeks after treatment | up to 8 weeks after first administration
  baseline-adjusted Oswestry Disability Index score at 8 weeks after treatment between study group(limaprost) and comparative group1(pregabalin) and combination group (limaprost + pregabalin)

SECONDARY OUTCOMES:
Initial Claudication Distance(ICD) on treadmill test | 4 and 8 weeks after first administration
  * Improvement of ICD at 4 weeks after first administration compared to baseline, between study group(limaprost) and comparative group1(pregabalin)
  * Improvement of ICD at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group 2(limaprost+ pregabalin)
lower extremity pain score measured by Visual Analog Scale(VAS) 10cm | 4 and 8 weeks after first administration
  * Change in VAS at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group1(pregabalin)
  * Change in VAS at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group 2(limaprost+ pregabalin)
Mean ratio of change in score of EuroQuol 5D (EQ-5D) | 4 and 8 weeks after first administration
  * Change in EQ-5D at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group1(pregabalin)
  * Change in EQ-5D at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group 2(limaprost+ pregabalin)
Mean ratio of change in score of Oswestry Disability Index(ODI) | 4 and 8 weeks after first administration
  * Change in ODI at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group1(pregabalin)
  * Change in ODI at 4, 8 weeks after first administration compared to baseline, between study group(limaprost) and comparative group 2(limaprost+ pregabalin)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hwan Moon, M.D.,Ph.D., Principal Investigator — Yonsei University College of Medicine Severance Hospital; Jin Hyok Kim, M.D.,Ph.D., Principal Investigator — Inje University; Jae Hyup Lee, M.D.,Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center; Suk Kyung Soo, M.D.,Ph.D., Principal Investigator — Kyunghee University Medical Center; Ho Joong Kim, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Ye Soo Park, M.D.,Ph.D., Principal Investigator — Hanyang University Guri Hospital; Moon Soo Park, M.D.,Ph.D., Principal Investigator — Hallym University Medical Center
Locations (7):
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Yonsei University Health System, Severance Hospital, Seoul, Seoul
  - KyungHee University Medical Center, Seoul, Seoul
  - Inje University Sanggye Paik Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul

REFERENCES:
- [Derived] Kim HJ, Kim JH, Park YS, Suk KS, Lee JH, Park MS, Moon SH. Comparative study of the efficacy of limaprost and pregabalin as single agents and in combination for the treatment of lumbar spinal stenosis: a prospective, double-blind, randomized controlled non-inferiority trial. Spine J. 2016 Jun;16(6):756-63. doi: 10.1016/j.spinee.2016.02.049. Epub 2016 Mar 29. PMID 27045252